CLINICAL TRIAL: NCT03385642
Title: Follow-Up Study Evaluating the Long-Term Outcomes of ChondroMimetic in the Treatment of Osteochondral Defects (Extension Study of Protocol 0MCM0107)
Brief Title: Follow-Up Study Evaluating the Long Term Outcome of ChondroMimetic in the Treatment of Osteochondral Defects in the Knee
Status: Completed | Type: Observational
Sponsor: Collagen Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: 0MCM0107-2
Record Dates: First submitted 2017-12-15; First posted 2017-12-28 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Osteochondral Defect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chondromimetic: Treatment of osteochondral defect in the knee with Chondromimetic device(s) in previous study 0MCM0107
  Interventions: Device: ChondroMimetic

INTERVENTIONS:
Device: ChondroMimetic — ChondroMimetic is a single-use, biphasic implant that serves as an osteochondral scaffold for the repair of cartilage defects in the knee

SUMMARY:
To investigate the long-term efficacy and safety of the medical device, ChondroMimetic, in subjects who were treated in the interventional study 0MCM0107 for osteochondral defects of the knee.

DETAILED DESCRIPTION:
This is an open-label, single center, extension study to the previous interventional study 0MCM0107 designed to investigate the long-term efficacy and safety of the medical device, ChondroMimetic, in the treatment of osteochondral defects of the knee. Follow-up to 6-months was completed as part of study 0MCM0107. All 17 subjects who received ChondroMimetic in study 0MCM0107 are eligible for enrolment into this extension study regardless of their current follow-up period.

ELIGIBILITY:
Treated with a Chondromimetic device under Protocol 0MCM0107 and completed the required follow-up.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects were treated with a Chondromimetic device under Protocol 0MCM0107
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Change from 0MCM0107 baseline in Modified Cincinnati Rating System | 0MCM0107 Baseline and through study completion, an average of approximately 8 years follow-up
  Subjective score designed to provide information regarding a patient's functional and clinical status after knee surgery.
KOOS (Knee injury and Osteoarthritis Outcome Score | Through study completion, an average of approximately 8 years follow-up
  Subjective score designed to provide information regarding a patient's functional and clinical status after knee surgery.
Cartilage repair tissue quantity and quality using 3D quantitative MRI analysis | Through study completion, an average of approximately 8 years follow-up
  Morphological segmentation utilizing a programmed anatomical atlas for all bone and cartilage structures will be used to assess defect filling (using previous MRI scans from study 0MCM0107 as reference), and T2 mapping for cartilage repair tissue quality.
Osteochondral defect repair assessment | Through study completion, an average of approximately 8 years follow-up
  Defect repair outcomes will be assessed using the magnetic resonance observation of cartilage repair tissue (MOCART) subjective radiological scoring system.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 0MCM0107 Baseline and through study completion, an average of approximately 8 years follow-up
  Long-term safety will be assessed by physical and knee examination, and subject history since original treatment in study 0MCM0107

CONTACTS AND LOCATIONS:
Overall Officials: Laszlo Hangody, MD, PhD, DSc, Principal Investigator — Uzsoki Hospital
Locations (1):
- Uzsoki Hospital, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No